CLINICAL TRIAL: NCT00814268
Title: COMbination of Clopidogrel and Aspirin for Prevention of REcurrence in Acute Atherothrombotic Stroke Study: Prospective, Randomized, Double-blind, Placebo-controlled, Multicenter Trial
Brief Title: COMbination of Clopidogrel and Aspirin for Prevention of Early REcurrence in Acute Atherothrombotic Stroke
Acronym: COMPRESS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLOPI_L_02452
Record Dates: First submitted 2008-12-23; First posted 2008-12-24 (Estimated); Last update posted 2014-02-28 (Estimated); Status verified 2014-02

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Clopidogrel; Aspirin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Combination therapy (Experimental): Administration of Aspirin + Clopidogrel for 30 days
  Interventions: Drug: Clopidogrel; Drug: Aspirin
- Monotherapy (Active Comparator): Administration of Aspirin + Clopidogrel placebo for 30 days
  Interventions: Drug: Clopidogrel placebo; Drug: Aspirin

INTERVENTIONS:
Drug: Clopidogrel — 75mg tablet, oral administration once daily
  Other Names: Plavix®
  Arms: Combination therapy
Drug: Clopidogrel placebo — Matching tablet, oral administration once daily
  Arms: Monotherapy
Drug: Aspirin — 100mg tablet, oral administration once daily

SUMMARY:
Primary objective:

* Comparison of efficacy of the combination therapy (clopidogrel plus aspirin) and the aspirin alone (main comparison) to prevent any recurrent ischemic lesion .

Secondary objectives:

* Comparison of Modified Rankin scale (mRS) scores;
* Comparison of the Incidence of all kinds of stroke and vascular death;
* Comparison of the Incidence of bleeding episodes (major and minor) and symptomatic intracerebral hemorrhages during the follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic stroke diagnosed within 48 hours from symptom onset;
* Cerebral ischemic lesion observed on diffusion-weighted magnetic resonance imaging (DWI MRI);
* Relevant atherothrombotic lesions on magnetic resonance angiography (MRA) or computed tomography angiography (CTA);
* Study drug administration within 48 hours from symptom onset;
* mRS score is 0-2 before the stroke.

Exclusion Criteria:

* Evidences of other relevant brain lesions such as Intracerebral hemorrhage (ICH) or brain tumor;
* Suspicious of stroke due to small-vessel occlusion;
* Stroke due to cardioembolism;
* Clinical necessity of conventional angiography or intervention before the end of study;
* Past history of ICH;
* Bleeding diathesis or coagulopathy;
* Chronic anemia (Hb<8.0) or thrombocytopenia (PLT<100K);
* Chronic liver disease (AST> 100 or ALT>100);
* Any other clinically relevant serious disease, including renal failure ( creatinine clearance<30mL/min);
* Allergy to Aspirin or clopidogrel;
* Subjected to intervention or surgical treatments within 3 months;
* Thrombolysis performed with rt-PA or UK after the stroke;
* Participation in another clinical study within the previous 30 days;
* Suspicious of poor drug compliance and requirements of the protocol;
* Females who are pregnant, breast-feeding, or childbearing potential and not using medically acceptable and effective contraception.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 358 (Actual)
Dates: Start 2008-12; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Number of participants with new ischemic lesions after the onset of acute atherothrombotic stroke | Within 30 days following the onset of acute atherothrombotic stroke

SECONDARY OUTCOMES:
Distribution of Modified Rankin Scale (mRS) scores | Day 30 after the onset of acute atherothrombotic stroke
Number of participants with non-fatal stroke, myocardial infarction (MI) or cardiovascular death (composite endpoint, first-ever) | Within 30 days following the onset of acute atherothrombotic stroke
Number of participants with stroke (all kinds) | Within 30 days following the onset of acute atherothrombotic stroke
Number of participants with bleeding episode (major or minor) | Within 30 days following the onset of acute atherothrombotic stroke
Number of participants with symptomatic intracerebral hemorrhage (ICH) | Within 30 days following the onset of acute atherothrombotic stroke

CONTACTS AND LOCATIONS:
Overall Officials: Hyang Rim Kim, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Seoul, South Korea

REFERENCES:
- [Derived] Hong KS, Lee SH, Kim EG, Cho KH, Chang DI, Rha JH, Bae HJ, Lee KB, Kim DE, Park JM, Kim HY, Cha JK, Yu KH, Lee YS, Lee SJ, Choi JC, Cho YJ, Kwon SU, Kim GM, Sohn SI, Park KY, Kang DW, Sohn CH, Lee J, Yoon BW; COMPRESS Investigators. Recurrent Ischemic Lesions After Acute Atherothrombotic Stroke: Clopidogrel Plus Aspirin Versus Aspirin Alone. Stroke. 2016 Sep;47(9):2323-30. doi: 10.1161/STROKEAHA.115.012293. Epub 2016 Jul 14. PMID 27418597